CLINICAL TRIAL: NCT04877587
Title: A Pilot Study of Gemcitabine Plus High-Dose Ascorbate in Locally Advanced Unresectable or Metastatic Soft Tissue and Bone Sarcomas Including Adolescents
Brief Title: Gemcitabine With Ascorbate Including Adolescents
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: David Dickens (Other)
Responsible Party: Sponsor-Investigator, David Dickens, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202009351
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma; Unresectable Soft Tissue Sarcoma; Metastatic Bone Sarcoma; Metastatic Soft-tissue Sarcoma; Unresectable Bone Sarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Ascorbic Acid; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ascorbate in combination with Gemcitabine (Experimental): The study will begin with a safety run-in.
  A patient-individualized pharmacokinetically-guided dose escalation design will be used for Ascorbate. Gemcitabine is administered following standard fixed dose infusion practice adopted at The University of Iowa Hospitals & Clinics. Ascorbate is infused prior to gemcitabine. Cycles are 28 days. Patients will be treated for a total of 6 cycles and assessed every 2 cycles for disease response.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbate — A patient-individualized pharmacokinetically-guided dose escalation design will be used for Ascorbate. The goal of the within-patient dose escalation is to achieve a target plasma ascorbate level between 20mM and 30mM. The administered dose levels under consideration are listed below.
  Dose Level Ascorbate
  * 2 60 g/m2 IV Days (1,2,8,9,15,16)
  * 1 50 g/m2 IV Days (1,2,8,9,15,16) 0 (Starting dose) 40 g/m2 IV Days (1,2,8,9,15,16)
    * 1 30 g/m2 IV Days (1,2,8,9,15,16)
  Other Names: Vitamin C
Drug: Gemcitabine — Gemcitabine 900 mg/m2 given at a fixed dose rate of 10 mg/m2/min on D1, D8 and D15 to be given over 90 min every 28 days
  Other Names: Gemzar®

SUMMARY:
The purpose of this research study is to see if a high dose of ascorbate (Vitamin C), in combination with the chemotherapy drug gemcitabine, is safe and effective in adolescents with locally advanced unresectable or metastatic soft tissue and bone sarcomas

DETAILED DESCRIPTION:
The primary objective of the expansion cohort of this pilot study is to evaluate preliminary evidence of anti-tumor activity of intravenous ascorbate in combination with gemcitabine as assessed by overall response rate to inform a subsequent Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 13 years to 17 years
* ECOG Performance Status of ≤ 2
* Ability to provide written informed consent from patient guardian and informed assent from patient; obtained prior to participation in the study and any related procedures being performed
* Tolerate a 10g ascorbate infusion (screening dose).
* Any patient with the diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except GIST and Kaposi's) from any site. A minimum of 1 prior chemotherapy regimen, including adjuvant or neo-adjuvant therapy for the treatment of sarcoma. Patients eligible for an anthracycline should have received a prior anthracycline containing regimen. Patients who decline or are not eligible for anthracycline treatment may be considered for this protocol as a first line treatment. Patients with a diagnosis of liposarcoma should also have received eribulin if they received anthracycline-based therapy prior to eribulin. Patients with a diagnosis of myxoid liposarcoma should have received trabectedin. Patients with angiosarcoma should have received either taxol or docetaxel. Patients must have measurable disease defined as at least 1 lesion ≥ 1cm in the greatest dimension.
* Patients with metastatic bone sarcomas who have failed all available therapies that have demonstrated clinical benefit. Available therapies include but not limited to methotrexate, adriamycin and cisplatin for osteosarcoma and vincristine, adriamycin and Cytoxan, ifosfamide, etoposide (VAC/IE) for Ewing's sarcoma.
* Previous exposure to Gemcitabine will only be allowed if there is no residual toxicity from previous treatments. Toxicity must be graded as 0 or 1 prior to study.
* Patients must have had disease progression on or following their most recent treatment regimen or on presentation for the first time with locally advanced unresectable or metastatic disease.

Exclusion Criteria:

Inadequate organ function as defined by:

Hematology:

* Neutrophil count of </=1,000/mm3
* Platelet count of </= 100,000/mm3L
* Hemoglobin < 9 g/dL (transfusion to meet eligibility allowed)

Biochemistry:

* AST/SGOT and ALT/SGPT >2.5 x upper limit of normal (ULN) or > 5.0 x ULN if the transaminase elevation is due to disease involvement
* Alkaline phosphatase >/=5 x ULN
* Serum bilirubin > 1.5 x ULN
* Serum creatinine > 1.5 x ULN or 24-hour creatinine clearance < 50 ml/min
* G6PD (glucose-6-phosphate dehydrogenase) deficiency
* Baseline MUGA or ECHO < than the lower limit of the institutional normal. ECHO or MUGA only done on patients with prior doxorubicin exposure.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Actively receiving insulin or requiring finger stick glucose monitoring at time of ascorbate infusion (unless an exception is granted by the IND sponsor, medical monitor, and the PI).
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Pregnancy (positive pregnancy test) or lactation.
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, warfarin and chlorpropamide. High dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs.
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy or any investigational drug < 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
* Concomitant use of any anti-cancer therapy or radiation therapy. Palliative radiation therapy to non-target lesions is permitted.
* Females of childbearing potential (FOCBP) who are unwilling to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
* Male patients whose sexual partners are FOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
* Patients with a history of another primary malignancy within 2 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs.37
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients with GIST tumors and Kaposi sarcoma are excluded
* Patients with history of more than one symptomatic oxalate stone in the last 6 months or visible stone in the kidney or ureter on screening CT scan.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events as defined by CTCAE version 5.0 | Adverse events will be followed for 4 weeks after the last pharmacologic ascorbate infusion
  Occurrence of adverse events as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number and severity of all adverse events will be summarized by simple descriptive statistics.
ORR as defined by RECIST 1.1 guidelines | For two years following completion of treatment
  Overall Response Rate (ORR) as defined by the percentage of patients with a complete or partial response, according to RECIST 1.1 guidelines

SECONDARY OUTCOMES:
PFS defined by RECIST 1.1 guidelines | For two years following completion of treatment
  Progression Free Survival (PFS) defined as the time from first day of study treatment to the first documented disease progression or death due to any cause, RECIST 1.1 guidelines
OS defined as the time from first day of study treatment to death due to any cause | For two years following completion of treatment
  Overall Survival (OS) defined as the time from first day of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: David Dickens, MD, FAAP, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No